CLINICAL TRIAL: NCT05739747
Title: Validation of the Gendolcat Score for the Prognosis of Chronic Postoperative Pain in Cesarean Section.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Consorci Sanitari de Terrassa (Other)
Responsible Party: Principal Investigator, Carles Espinos Ramírez, M.D., Consorci Sanitari de Terrassa
Other Study IDs: 02-23-270-003
Record Dates: First submitted 2023-02-05; First posted 2023-02-22 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Chronic Post Surgical Pain; Cesarean Section Complications; Chronic Pain
MeSH Terms: conditions — Pain, Postoperative; Chronic Pain | interventions — Surveys and Questionnaires; Restraint, Physical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women undergoing cesarean section: This study is designed with a single cohort of women who will undergo a scheduled cesarean section
  Interventions: Other: Questionnaire; Other: Questionnaire via telephone call; Other: Physical examination

INTERVENTIONS:
Other: Questionnaire — All patients should complete the following questionnaires:
  On the day of surgery:
  * Patient registration.
  * Complete medical history.
  * Gendolcat scale (including the Spanish version of the SF-12 scale).
  * Spanish version of the catastrophizing scale.
Other: Questionnaire — The investigators should complete a questionnaire during the surgical procedure specifying the anesthetic technique used, drugs and doses used and record any incident during the surgical procedure
Other: Questionnaire — The investigators should complete a questionnaire 24 hours after surgery to assess the possible presence of postoperative pain as well as the intensity and need for rescue analgesia.
Other: Questionnaire via telephone call — At 3 months, patients will be called and a structured questionnaire will be completed to assess the presence of chronic postoperative pain.
Other: Physical examination — Those women who, after the telephone call, are considered to have chronic post-surgical pain will undergo a physical examination to confirm it. The type of pain and its intensity will also be evaluated. The impact on their daily physical activity and quality of life will be evaluated by means of a questionnaire.

SUMMARY:
Chronic post-surgical pain is a problem that has historically been underestimated. Over the last few years there has been a search for strategies to both predict and prevent its occurrence in patients undergoing surgery. The Gendolcat index is the only predictive model that uses only objective pre-surgical variables to assess the risk of suffering chronic post-surgical pain. However, it is only validated for the following surgeries: thoracotomy, hysterectomy and open inguinal hernia. Our aim is to test whether the Gendolcat model is also valid for cesarean section.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent elective caesarean section.
* Patients who have previously signed the informed consent form.

Exclusion Criteria

* Urgent cesarean section.
* Patients with severe psychiatric pathology.
* Patients who require a different surgical approach than usual.
* Patients who refuse to take part in the study and/or to sign the informed consent form.

informed consent.

- Patients with a high language barrier.

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Patients undergoing elective cesarean section.
Sampling Method: Non-Probability Sample
Enrollment: 371 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-02 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Gendolcat score | The Gendolcat score will be assessed on the day patients are included in the study
  The Gendolcat score assesses the likelihood of suffering chronic post-surgical pain
Categoric Pain Scale | Done during physical examination will be performed 3 months after cesarean section.
  These pain scales give people a simple way to rate their pain intensity using a verbal or visual descriptor of their pain.
Numeric Pain Scale | Done during physical examination will be performed 3 months after cesarean section.
  Patients are asked to circle the number between 0 and 10, 0 and 20 or 0 and 100 that fits best to their pain intensity
Short Edition of the Brief Pain Inventory | Done during physical examination will be performed 3 months after cesarean section.
  Rapidly assesses the severity of pain and its impact on functioning
DN4 Questionnaire | Done during physical examination will be performed 3 months after cesarean section.
  To estimate the probability of neuropathic pain

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schug SA, Lavand'homme P, Barke A, Korwisi B, Rief W, Treede RD; IASP Taskforce for the Classification of Chronic Pain. The IASP classification of chronic pain for ICD-11: chronic postsurgical or posttraumatic pain. Pain. 2019 Jan;160(1):45-52. doi: 10.1097/j.pain.0000000000001413. PMID 30586070
- [Background] Kehlet H, Jensen TS, Woolf CJ. Persistent postsurgical pain: risk factors and prevention. Lancet. 2006 May 13;367(9522):1618-25. doi: 10.1016/S0140-6736(06)68700-X. PMID 16698416
- [Background] Stuart AR, Kuck K, Naik BI, Saager L, Pace NL, Domino KB, Posner KL, Alpert SB, Kheterpal S, Sinha AK, Brummett CM, Durieux ME; the MPOG EOS Investigator Group. Multicenter Perioperative Outcomes Group Enhanced Observation Study Postoperative Pain Profiles, Analgesic Use, and Transition to Chronic Pain and Excessive and Prolonged Opioid Use Patterns Methodology. Anesth Analg. 2020 Jun;130(6):1702-1708. doi: 10.1213/ANE.0000000000004568. PMID 31986126
- [Background] Althaus A, Hinrichs-Rocker A, Chapman R, Arranz Becker O, Lefering R, Simanski C, Weber F, Moser KH, Joppich R, Trojan S, Gutzeit N, Neugebauer E. Development of a risk index for the prediction of chronic post-surgical pain. Eur J Pain. 2012 Jul;16(6):901-10. doi: 10.1002/j.1532-2149.2011.00090.x. Epub 2011 Dec 23. PMID 22337572
- [Background] Mathes T, Pape-Kohler C, Moerders L, Lux E, Neugebauer EAM. External Validation and Update of the RICP-A Multivariate Model to Predict Chronic Postoperative Pain. Pain Med. 2018 Aug 1;19(8):1674-1682. doi: 10.1093/pm/pnx242. PMID 29121211
- [Background] Meretoja TJ, Andersen KG, Bruce J, Haasio L, Sipila R, Scott NW, Ripatti S, Kehlet H, Kalso E. Clinical Prediction Model and Tool for Assessing Risk of Persistent Pain After Breast Cancer Surgery. J Clin Oncol. 2017 May 20;35(15):1660-1667. doi: 10.1200/JCO.2016.70.3413. Epub 2017 Mar 13. PMID 28524782
- [Background] Montes A, Roca G, Cantillo J, Sabate S; GENDOLCAT Study Group. Presurgical risk model for chronic postsurgical pain based on 6 clinical predictors: a prospective external validation. Pain. 2020 Nov;161(11):2611-2618. doi: 10.1097/j.pain.0000000000001945. PMID 32541391
- [Background] Montes A, Roca G, Sabate S, Lao JI, Navarro A, Cantillo J, Canet J; GENDOLCAT Study Group. Genetic and Clinical Factors Associated with Chronic Postsurgical Pain after Hernia Repair, Hysterectomy, and Thoracotomy: A Two-year Multicenter Cohort Study. Anesthesiology. 2015 May;122(5):1123-41. doi: 10.1097/ALN.0000000000000611. PMID 25985024
- [Background] Nikolajsen L, Sorensen HC, Jensen TS, Kehlet H. Chronic pain following Caesarean section. Acta Anaesthesiol Scand. 2004 Jan;48(1):111-6. doi: 10.1111/j.1399-6576.2004.00271.x. PMID 14674981
- [Background] Jin J, Peng L, Chen Q, Zhang D, Ren L, Qin P, Min S. Prevalence and risk factors for chronic pain following cesarean section: a prospective study. BMC Anesthesiol. 2016 Oct 18;16(1):99. doi: 10.1186/s12871-016-0270-6. PMID 27756207
- [Background] Sharma LR, Schaldemose EL, Alaverdyan H, Nikolajsen L, Chen D, Bhanvadia S, Komen H, Yaeger L, Haroutounian S. Perioperative factors associated with persistent postsurgical pain after hysterectomy, cesarean section, prostatectomy, and donor nephrectomy: a systematic review and meta-analysis. Pain. 2022 Mar 1;163(3):425-435. doi: 10.1097/j.pain.0000000000002361. PMID 34121077